CLINICAL TRIAL: NCT07337590
Title: Anastomotic Safety and Surveillance Using Real-time Enhanced Sensing Using xBar
Acronym: ASSURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Exero Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP 04
Record Dates: First submitted 2025-12-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will include two cohorts:
  * Interventional Cohort: Approximately 80 eligible subjects with colorectal cancer undergoing elective low anterior resection with anastomosis, without concomitant diversion, who meet all study inclusion criteria and none of the exclusion criteria.
  * Historical Control Cohort: A de-identified historical cohort consisting of a matched population that underwent surgical procedures during 2023. Historical data will include subject demographics, initial diagnosis, index surgery details, tumor location, comorbidities, length of stay (LOS), and readmission rates following the index colorectal surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Interventional Cohort (Experimental): The xBar drain will be placed during the elective low anterior resection, which will be performed according to each medical center's standard surgical procedures. Following placement, the xBar system will continuously collect measurements until drain removal.
  Interventions: Device: xBar™ System
- Historical Control Cohort (No Intervention): A de-identified historical cohort consisting of a matched population that underwent surgical procedures during 2023. Historical data will include subject demographics, initial diagnosis, index surgery details, tumor location, comorbidities, length of stay (LOS), and readmission rates following the index colorectal surgery.

INTERVENTIONS:
Device: xBar™ System — Device: The xBar™ device functions by integrating a sensing electrode array into a standard surgical drain, thereby enabling monitoring without altering standard surgical protocols Description: The Exero Medical xBar™ System is designed to provide continuous postoperative monitoring of gastrointestinal (GI) anastomoses to support the early identification of anastomotic leaks. The device functions by integrating a sensing electrode array into a standard surgical drain, thereby enabling monitoring without altering standard surgical protocols.
  Arms: Interventional Cohort

SUMMARY:
Purpose: To evaluate the effect of xBar system utilization on clinical outcomes during recovery following colorectal surgery.

DETAILED DESCRIPTION:
The study is intended to evaluate the effect of xBar utilization on clinical outcomes during recovery from colorectal surgery. During the study, patients in the intervention group admitted for low anterior resection surgery will have xBar placed during their index surgery. The overall morbidity, healthcare utilization costs, and stoma utilization of the intervention group will be compared to those of the historical control group, consisting of patients meeting the same inclusion/exclusion criteria of the patients in the intervention group.

The xBar system, classified as a non-significant risk device in the pivotal study, is designed as an integrated platform for post-operative monitoring, built to fit into the existing clinical workflow without altering the standard surgical protocol.

ELIGIBILITY:
Inclusion Criteria:

Interventional Cohort

1. Adults (≥21 years) scheduled for elective low anterior resection (by any surgical technique), due to colorectal cancer
2. Expected anastomosis within 10 cm from the anal verge
3. Usage of drain during the surgery (to be confirmed during the surgery)
4. Willing and able to comply with the study follow up and able and agree to provide informed consent.

Historical Cohort

1. Adults aged ≥21 years at the time of surgery.
2. Underwent a low anterior resection (LAR) for malignant colorectal disease.
3. Documented colorectal anastomosis located <10cm from the anal verge, or documented tumor <10cm from the anal verge. Complete documentation for the index hospitalization and for the required 12-month follow-up period, or up to stoma take down procedure whichever came first.

Exclusion Criteria:

Interventional Cohort

1. Subjects with benign disease
2. Contraindication for surgery and/or general anesthesia.
3. Known pregnancy or lactation.
4. Subjects receiving prophylactic stoma formation during index surgery (to be confirmed intraoperatively)
5. Known electronic devices implanted in the chest or the abdominal cavity (e.g., pacemaker, cardioverter/defibrillator).
6. Major medical or psychiatric illness or condition, or other factors that may affect general health or ability to adhere to the follow-up schedule.
7. Known allergic reactions to materials used in the components of the xBar system, i.e., silicone, rubber and stainless-steel.
8. Participation in another interventional study during the xBar system usage. Historical Cohort

1. LAR performed for benign or non-oncologic indications (e.g., diverticulitis, inflammatory bowel disease, non-malignant strictures, fistula).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint-Demonstrate non-inferiority between the study interventional and historical cohorts | At the time points of 30 and 90 days following index surgery
  Non-inferiority of the mean Modified Comprehensive Complication Index (MCCI) of the modified intent-to-treat (mITT) population at 30 days following the index surgery, compared with the MCCI of the matched historical cohort.
Primary Safety Endpoint - No Unexpected Serious Adverse Device Events within the Intent to Treat population during the study period ( up to 365 days following index surgery) | from the date of index surgery up to 365 days following the index surgery
  Lack of unanticipated serious adverse events related to the xBar system or xBar procedure during the study period ( up to 365 days from the index surgery)

SECONDARY OUTCOMES:
Number of Stoma-Free patients during the study follow up | Time points 30 days, 90 days, 6 months and 12 months following the index surgery
  Comparison of the number of stoma-free patients in the intervention group vs. the historical cohort at postoperative day 30, postoperative day 90, 6 months, and 12 months. (in %)
Sensitivity and specificity of xBar outcome | As from Visit 0 (Day of Surgery -drain placement) through the discharge visits (drain removal as per routine practice), anticipated average 3 days.
  Evaluation of xBar's leak detection performance (Sensitivity, Specificity, Negative Predictive Value, Positive Predictive Value).
1. Comparison of MCCI Comorbidity Index (between study cohorts) 2. Number of Stome-Free patients during the study follow up 3. Sensitivity and specificity of xBar outcome | At timepoints of 30, 90 ,180 and 365 days following the index surgery
  1. Comparison of MCCI (Comorbidity Index) score based on National Surgical Quality Improvement Program scores, length of stay and readmission events at postoperative day 30 in the intervention group VS the historical cohort
  2. Comparison of percentages of stoma-free patients in the intervention group vs. the historical cohort at POD30, POD90, 6 months, and 12 months.
  3. Evaluation of xBar's leak detection performance (Sensitivity, Specificity, Negative Predictive Value, Positive Predictive Value).

OTHER OUTCOMES:
Tertiary Endpoint- Health Resource Utilization | Post operative days 30, 90 and 6 months, 12 months
  Comparative assessment between study cohorts of overall and specific healthcare resource utilization related to index surgery and postoperative recovery at post operative days 30, 90 and 6 months, 12 months.
Exploratory Endpoint-Clinical Teams Usability Feedback | As from Visit 0 (Day of Surgery -drain placement) through the discharge visits (drain removal as per routine practice), anticipated average 3 days.]
  Use of questionnaires to collect feedback from clinical teams on system setup, intraoperative integration, postoperative monitoring, and decision-support utility.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Louisville Hospital, Louisville, Kentucky
  - Weill Cornell Medicine Colon and Rectal Surgery, New York, New York
  - Department of Colon and Rectal Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No